CLINICAL TRIAL: NCT05738642
Title: Evaluation of the Efficacy of Early Bunching of a Four-factor Prothrombin Complex Concentrates in Patients With Severe Traumatic Hemorrhage: a Multicenter, Randomized Controlled, Open-label Clinical Study
Brief Title: Evaluation of the Efficacy of Early Bunching of a FF-PCC in Patients With Severe Traumatic Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0955
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Trauma
Keywords: trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4F-PCC group (Experimental): 1. Basic and normative treatment in accordance with the European Guidelines for Major Bleeding 2019: effective hemostatic measures and target-oriented correction of coagulation function. 2. 4 F- PCC by intravenous infusion of cluster
  Interventions: Drug: 4 factor Prothrombin Complex Concentrates
- non 4F-PCC group (No Intervention): 1. Basic and normative treatment in accordance with the European Guidelines for Major Bleeding 2019: effective hemostatic measures and target-oriented correction of coagulation function.

INTERVENTIONS:
Drug: 4 factor Prothrombin Complex Concentrates — Cluster 4 f - PCC by intravenous infusion (boya 4 f - PCC, a bottle of 400 IU) : 25 IU/kg dose infusion time: as soon as possible after admission infusion, at the latest within 2 hours after admission to infusion infusion method: Sodium chloride injection 5% glucose injection was diluted into 50 ml per bottle, and then intravenous infusion was carried out with a blood transfusion device with a mesh device. The infusion was finished in 60-120 minutes
  Other Names: test group
  Arms: 4F-PCC group

SUMMARY:
Uncontrolled hemorrhage within 24 hours after severe trauma is the main cause of death in trauma patients. Hemorrhagic shock may be accompanied by traumatic coagulopathy in the early stages of severe trauma. Among them, the main pathogenesis of traumatic coagulation disorder is tissue injury, hypoperfusion, inflammatory response and acute neurohumoral system activation leading to the activation of endogenous protein C, increased consumption of coagulation factor, loss of coagulation factor caused by massive bleeding, low temperature and other factors aggravate the disorder of coagulation function and cause hyperfibrinolysis. Studies have shown that the fatality rate of patients with severe traumatic coagulopathy is 4-8 times higher than that of patients without coagulopathy. Active and effective injury-controlled resuscitation and surgical treatment, target-oriented supplementation of coagulation substrate and correction of coagulation function are the main measures for high-quality treatment of patients with severe trauma. Therefore, early improvement of coagulation function is the key to improve the comprehensive treatment level of patients with severe trauma.

At present, four-factor prothrombin complex (4F-PCC) is a compound preparation containing coagulation factors Ⅱ, VII, IX and X separated from fresh plasma of healthy people. It is used in clinical treatment of patients with coagulation factor deficiency or bleeding complicated by taking anticoagulant drugs to achieve rapid hemostasis effect. However, large-scale, long-term observation of the efficacy and safety of the early application of cluster infusion of 4F-PCC in traumatic massive hemorrhage, correction of cocoagulation dysfunction, and improvement of clinical prognosis has not been proven.

This study intends to conduct a clinical intervention study on early bunching and sufficient use of 4F-PCC in patients with severe traumatic massive hemorrhage, and evaluate its efficacy in early use of severe traumatic massive hemorrhage through a randomized controlled and open-label clinical study of multi-center, bunching use of PCC in patients with severe traumatic massive hemorrhage.

DETAILED DESCRIPTION:
Trauma causes at least 5.8 million deaths globally every year, accounting for 1/10 of the global annual death toll [1, 2]. Uncontrolled bleeding within 24h after trauma is the main cause of death in trauma patients [3, 4], and about 1/3 patients are accompanied by traumatic coagulopathy upon admission [5, 6]. Studies and analyses have shown that fatal traumatic hemorrhage is the most common preventable death factor [7]. The implementation of early deterministic and effective hemostatic measures for patients with severe traumatic massive hemorrhage can significantly reduce clinical massive hemorrhage and timely correct hemorrhagic shock, and it is necessary to correct traumatic coagulopathy and other traumatic complications [8, 9]. The occurrence of traumatic coagulopathy is caused by multiple factors, including severe tissue trauma and hypoperfusion drive, traumatic blood loss, massive intravenous infusion of hypocoagulable blood products such as crystal solution or red blood cells resulting in blood dilution, acidosis, depletion of coagulation factors, and even hypothermia and excessive inflammation can lead to the exacerbation of coagulopathy. Patients with systemic hypocoagulation and hyperfibrinolysis. In addition, traumatic coagulopathy, as one of the "death triad" of severe trauma, is associated with the increased need for hospitalization blood transfusion, prolonged mechanical ventilation, multiple organ failure and other increased risk of trauma complications. In addition, the fatality rate of trauma patients with severe traumatic coagulodysfunction is 4-8 times higher than that of patients without severe traumatic coagulodysfunction [5, 10, 11]. Therefore, for patients with severe traumatic hemorrhage complicated with coagulopathy, positive values should be adopted to rapidly improve the coagulopathy of patients and improve clinical prognosis.

The treatment of severe traumatic hemorrhage, hemorrhagic shock and traumatic coagulopathy includes timely correction of massive hemorrhage, timely use of proportional transfusion of blood products to ensure effective fluid volume resuscitation and temperature maintenance, and achieve target-oriented correction of coagulopathy while taking into account thrombosis prevention and other comprehensive therapeutic strategies [12]. Among them, proportional infusion of RBC and Fresh Frozen Plasma (FFP) in clinical mass transfusion protocol (MTP) is still the most commonly used therapeutic measure [13, 14]. However, with the increasing imbalance between supply and demand of blood products, some treatment units often face the dilemma of lack of blood products. Therefore, more and more European and American countries begin to apply Coagulation Factor Concentrates (Coagulation Factor Concentrates, CFCs) included Prothrombin Complex Concentrates (PCC) and Fibrinogen Concentrates (FC) for early resuscitation and target-directed coagulation management. Compared with FFP alone, the advantages of CFCs to correct coagulation dysfunction include: by providing standardized and high concentration of coagulation factors, reducing virus transmission and transfusion-related adverse reactions (such as acute respiratory distress syndrome, sepsis and multiple organ failure), immediate use without matching, and easy operation [15, 16]; The bunching of PCCS can effectively reduce the need for blood transfusion, achieve faster correction of coagulation function and reduce in-hospital mortality [12, 17-19]. A prospective, single-center, randomized controlled trial found that early use of fibrinogen concentrate (FC) may reduce blood transfusion volume and the incidence of multiple organ failure [17]. However, at present, for patients with severe trauma and massive hemorrhage, the use of MTP and blood products can only be effectively implemented on the basis of the completion of coagulation function test, accurate thrombus elastogram (TEG) and dynamic evaluation of the body's coagulation function [12, 17]. However, the acquisition of TEG test results is often slow, which cannot timely and effectively guide clinicians to carry out target-oriented use of blood products and clinical mass transfusion in early stage. In addition, when hemorrhagic shock cannot be effectively corrected in patients with severe traumatic massive hemorrhage in the early stage, timely treatment of coagulopathy is delayed. In conclusion, timely and sufficient supplement of prothrombin complex PCC and other blood products may have certain application value for timely and effective correction of coagulation dysfunction.

Prothrombin complex (PCC) is a kind of plasma protein concentrate containing coagulation factor which is isolated and prepared from healthy human mixed plasma. Currently, there are two types of clinically available PCCS: 3-factor prothrombin complex (3F-PCC) and 4-factor prothrombin complex (4F-PCC) [20]. 4F-PCC is a compound preparation containing coagulation factor Ⅱ, VII, IX and X, which has been used in clinical treatment of patients with coagulation factor deficiency or bleeding complicated by taking anticoagulant drugs to achieve rapid hemostatic effect. Studies have shown that compared with 3F-PCC, 4F-PCC can better reduce mortality and treatment costs in the management of traumatic coagulopathy [21]. However, the efficacy and safety of 4F-PCC in early dosing and bunching of traumatic massive bleeding have not been demonstrated by prospective multicenter randomized controlled trials. In addition to the application of PCC in patients with traumatic hemorrhage complicated by anticoagulant drugs, the European Guidelines for Massive Hemorrhage 2019 Edition lacks clear guidelines for the treatment of patients with severe traumatic hemorrhage complicated with coagulopathy. Nevertheless, there is widespread clinical concern that PCCS increase the risk of thromboembolic complications; In trauma patients, retrospective studies have shown that the incidence of different thrombus varies from 2% to 15% [17, 19, 22]. A previous retrospective study in the hospital where the author worked showed that 17.5% of severe trauma patients used 4F-PCC empirically, and the incidence of thrombosis and other adverse events in these patients was about 3%. Since the late 1990s, in order to improve safety, activators have been removed and anticoagulant factors added to most PCC processes to balance the risk of thrombotic complications [23]. In vitro studies of severe trauma have also found that appropriate doses of 4F-PCC can safely improve coagulation function and reduce blood loss [24], and the thrombotic potential of 4F-PCC is lower than that of aPCC or rFVIIa [25]. Pharmacovigilance data suggest that the risk of thromboembolic complications in PCC may be low, but the primary source of these data is vitamin K antagonist reversal [26]. Therefore, for the application of PCC in the management of traumatic coagulopathy, there is still a lack of scientific clinical practice guidance basis, and systematic prospective research is needed at the same time.

We noted that two large randomized controlled trials were registered in ClinicalTrials.gov by European and American teams. One was the combination of PCC+FC administration in patients with traumatic bleeding, and the other was the use of PCC alone, but both trials did not take reduction of transfusion of blood products as the main evaluation index [20, 27, 28]. It is worth mentioning that a recently published meta-analysis of retrospective studies found that the use of PCCS was associated with reduced mortality in trauma patients [29]. Therefore, we can assume that early use of 4F-PCC in severe trauma with hemorrhagic shock can correct bleeding and coagulodysfunction as soon as possible, thereby preventing circulatory, respiratory and renal multiple organ failure and improving prognosis. In addition, the lack of blood products and the difficulty in the implementation of massive blood transfusion plan also put forward a higher demand for the early and efficient use of clotting substrates in the treatment of patients with massive traumatic hemorrhage. This has also become an important research content in this study, such as the early empirical use of 4-PCC to improve the clinical prognosis of patients with severe traumatic massive hemorrhage, reduce the need for blood products, quickly correct coagulation dysfunction, and reduce the risk of thrombosis events. Therefore, this study intends to conduct early empirical bunching of 4-PCC in patients with severe traumatic massive hemorrhage, and evaluate its effectiveness and safety in the early stage of severe traumatic massive hemorrhage through a multicenter, randomized controlled, open-label study. To further improve the treatment of traumatic massive hemorrhage to provide a certain reference basis; It also provides the theoretical basis and clinical practice for correcting coagulation dysfunction in the early stage of severe trauma treatment.

ELIGIBILITY:
Inclusion Criteria:

(1) The age of adult trauma patients ≥18 years, < The 80 - year - old (2) ISS> 16 (3) emergency preview class for 1 to 2; (4) after trauma & lt; 3 hours; Trauma induced active bleeding; (5) blood consumption (ABC) score of 2 or more, or a preliminary assessment of blood loss & gt; 1000ml or ≥4 units of red blood cells expected to be transfused

Exclusion Criteria:

(1) history of anticoagulation and antiplatelet drugs (2) has a deep venous thromboembolism (VTE) and pulmonary embolism (PE) history (3) (4) on patients with severe head injury occurred cardiac arrest patients (5) lactation, pregnant women 6 Abdominal cavity viscera perforation surgical treatment in patients with 7) in patients with sepsis shock patients with all kinds of mental illness incapacitated pet-name ruby are unknown agent for informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of multiple organ failure within 7 days | 7 days
mortality at 28 days | 28 days

SECONDARY OUTCOMES:
The total transfusion volume of blood products within 24 hours after trauma | 28 days
  The total transfusion volume of blood products within 24 hours after trauma

CONTACTS AND LOCATIONS:
Overall Officials: yongan xu, doctor, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University